CLINICAL TRIAL: NCT04570930
Title: Improving Outcomes for Care Partners of Persons With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Noelle E Carlozzi, Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00181282; 2R01NR013658 (NIH)
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Caregivers
Keywords: Stress; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This behavioral trial will use a 2-arm randomized controlled design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Just-in-time adaptive intervention (JITAI) (Experimental): Participants will wear the Fitbit®, provide daily reports of Health- Related Quality of Life (HRQOL) and receive personalized pushes over a six-month (180 day) period.
  Interventions: Behavioral: Just-in-time adaptive intervention (JITAI)
- Control (Active Comparator): Participants will wear the Fitbit® and provide daily reports of HRQOL over a six-month (180 day) period (without the personalized feedback).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Just-in-time adaptive intervention (JITAI) — JITAI is an emerging intervention that incorporates passive mobile sensor data feedback (sleep and activity [step] data from a Fitbit ®), and real-time self-reporting of HRQOL via a study specific app called CareQOL to provide personalized feedback via app alert.
  Arms: Just-in-time adaptive intervention (JITAI)
Behavioral: Control — Participants will wear the Fitbit® and provide daily reports of HRQOL over a six-month (180 day) period.
  Arms: Control

SUMMARY:
Care partners of persons with traumatic brain injury (TBI) are often faced with considerable physical and emotional stress resulting from their caregiver role. The researchers hypothesize that the care partners who receive the intervention will show improvements in caregiver strain and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Be caring for an adult (age 18 or above) with a medically documented TBI that is ≥1-year post-injury and meets the TBI Model Systems (TBIMS) criteria for complicated mild, moderate or severe TBI and who sustained their TBI at age 16 or older
* Provide emotional, physical, and/or financial support/assistance to the individual with the TBI, indicating a response ≥1 to the following question: "On a scale of 0-10, where 0 is "no assistance" and 10 is "assistance with all activities", how much assistance does the person you care for require from you to complete activities of daily living due to problems resulting from his/her TBI? Activities could consist of personal hygiene, dressing and undressing, housework, taking medications, managing money, running errands, shopping for groceries or clothing, transportation, meal preparation and cleanup, remembering things, etc."
* Have access to necessary resources for participating in a technology-based intervention (smartphone/tablet and internet access) and be willing to use their personal equipment/internet for this study, including downloading the study app and the Fitbit® app on their mobile device
* Is able and willing to complete all study assessments for the duration of their study participation (approximately 375 days)

Exclusion Criteria:

* Is a professional, paid caregiver (e.g., home health aide)
* Anything that would preclude safe or meaningful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Carlozzi, Ph.D., Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Participant data collected during the trial, after de-identification, will be available for sharing with individuals in the scientific community, upon request. The data will be available after the acceptance for publication of the main findings from the final dataset. The University of Michigan Project Manager will coordinate requests for data and maintain documentation for requests and distributions. An institutional data use agreement will be required before data is shared.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available after the acceptance for publication of the main findings from the final dataset.
Access Criteria: Data is available upon request to the project manager. Requests for data sharing should be emailed to PMR-CODAlab@med.umich.edu

REFERENCES:
- [Derived] Carlozzi NE, Choi SW, Wu Z, Sen S, Troost J, Lyden AK, Miner JA, Graves C, Sander AM. The reliability and validity of the TBI-CareQOL system in four diverse caregiver groups. J Patient Rep Outcomes. 2023 Jun 26;7(1):57. doi: 10.1186/s41687-023-00602-x. PMID 37358716
- [Derived] Carlozzi NE, Sander AM, Choi SW, Wu Z, Miner JA, Lyden AK, Graves C, Sen S. Improving outcomes for care partners of persons with traumatic brain injury: Protocol for a randomized control trial of a just-in-time-adaptive self-management intervention. PLoS One. 2022 Jun 9;17(6):e0268726. doi: 10.1371/journal.pone.0268726. eCollection 2022. PMID 35679283

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Just-in-time Adaptive Intervention (JITAI) | Control
Started | 129 | 128
Completed | 122 | 122
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Just-in-time Adaptive Intervention (JITAI) | Control | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (15.3) | 52 (14.3) | 52 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 103 | 204
  Male | 28 | 25 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 19 | 41
  Not Hispanic or Latino | 107 | 109 | 216
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 20 | 16 | 36
  White | 98 | 100 | 198
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 129 | 128 | 257
Self-reported Caregiver Strain Measured by Traumatic Brain Injury Caregiver Quality of Life [Mean (Standard Deviation); unit: T-score] — TBI-CareQOL Caregiver Strain assesses perceived feelings of feeling overwhelmed, stressed and "beat-down" related to the care partner role. Self-reported responses are on a Likert scale. The measure is scored on a T metric with a mean of 50 and a standard deviation of 10. Higher scores indicate more strain.
  T-score | 51.0 (8.2) | 49.3 (8.6) | 50.1 (8.4)
Self-reported Anxiety Score Measured by Patient-Reported Outcomes Measurement Information System [Mean (Standard Deviation); unit: T-score] — PROMIS Anxiety assesses self-reported feelings of fear, anxiety and hyper-arousal. Self-reported responses are on a Likert scale. The measure is scored on a T metric with a mean of 50 and a standard deviation of 10. Higher scores indicate more anxiety.
  T-score | 57.5 (7.1) | 56.1 (9.3) | 56.8 (8.3)
Self-reported Depression Score Measured by Patient-Reported Outcomes Measurement Information System [Mean (Standard Deviation); unit: T-score] — PROMIS Depression assesses self-reported feelings of sadness and worthlessness. Self-reported responses are on a Likert scale. The measure is scored on a T metric with a mean of 50 and a standard deviation of 10. Higher scores indicate more depression.
  T-score | 53.5 (7.3) | 53.0 (8.6) | 53.3 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Self-reported Caregiver Strain as Measured by Traumatic Brain Injury Caregiver Quality of Life (TBI-CareQOL) Caregiver Strain
Description: TBI-CareQOL Caregiver Strain assesses perceived feelings of feeling overwhelmed, stressed and "beat-down" related to the care partner role. Self-reported responses are on a Likert scale. The measure is scored on a T metric with a mean of 50 and a standard deviation of 10. Higher scores indicate more strain.
Time Frame: Baseline, Day 180 of intervention
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Just-in-time Adaptive Intervention (JITAI) | Control
Number analyzed (Participants) | 122 | 122
T Score | -1.09 (7.76) | 0.34 (6.53)

2. Secondary Outcome: Change From Baseline in Self-reported Anxiety Score as Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety
Description: PROMIS Anxiety assesses self-reported feelings of fear, anxiety and hyper-arousal. Self-reported responses are on a Likert scale. The measure is scored on a T metric with a mean of 50 and a standard deviation of 10. Higher scores indicate more anxiety.
Time Frame: Baseline, Day 180 of intervention
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Just-in-time Adaptive Intervention (JITAI) | Control
Number analyzed (Participants) | 122 | 122
T Score | -1.14 (7.58) | 0.60 (8.23)

3. Secondary Outcome: Change From Baseline in Self-reported Depression Score as Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Depression
Description: PROMIS Depression assesses self-reported feelings of sadness and worthlessness. Self-reported responses are on a Likert scale. The measure is scored on a T metric with a mean of 50 and a standard deviation of 10. Higher scores indicate more depression.
Time Frame: Baseline, Day 180 of intervention
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Just-in-time Adaptive Intervention (JITAI) | Control
Number analyzed (Participants) | 122 | 122
T Score | -1.01 (7.12) | 0.61 (7.75)

ADVERSE EVENTS:
Time Frame: Baseline to Day 360
Arm/Group | Just-in-time Adaptive Intervention (JITAI) | Control
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/128
Serious Adverse Events (participants affected / at risk) | 1/129 | 1/128
Other Adverse Events (participants affected / at risk) | 17/129 | 32/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Just-in-time Adaptive Intervention (JITAI) (N=129) | Control (N=128)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) — Participant was hospitalized for COVID-19.
Pancreatitis (Endocrine disorders) | 0 | 1 (3) — Participant reported flares of pancreatitis and reported 3 admissions to the hospital.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Just-in-time Adaptive Intervention (JITAI) (N=129) | Control (N=128)
COVID-19 (Infections and infestations) | 6 (6) | 9 (9)
Skin irritation from Fitbit wristband (Skin and subcutaneous tissue disorders) | 7 (8) | 10 (10) — Skin irritation including itching or rash
Increased mental health problems (Social circumstances) | 9 (13) | 15 (22) — Participant reported increase in mental health symptoms including increased stress, depression, or anxiety

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04570930/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT04570930/ICF_001.pdf